CLINICAL TRIAL: NCT02480985
Title: Clinical Outcomes and Predictors of PITuitary Disorders in Patients With Moderate and Severe Traumatic Brain Injury: the PIT-TBI Prospective Multicenter Pilot Cohort Study
Brief Title: The PIT-TBI Pilot Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: CHU de Quebec-Universite Laval (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Canadian Critical Care Trials Group (Other); Fonds de la Recherche en Santé du Québec (Other Government)
Responsible Party: Principal Investigator, François Lauzier, MD MSc FRCPC, CHU de Quebec-Universite Laval
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: C14-06-2040-21
Record Dates: First submitted 2015-06-18; First posted 2015-06-25 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Pituitary Disorders; Traumatic Brain Injury
Keywords: Pituitary Disorders; Traumatic Brain Injury; Critical Care; Outcome Research; Risk Factors; Patient Oriented Research
MeSH Terms: conditions — Pituitary Diseases; Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pituitary function evaluation (Other): Exams performed according to a determined schedule following admission in the intensive care unit in order to determine the risk factors and the outcome associated with pituitary disorders.
  Interventions: Other: Pituitary function evaluation

INTERVENTIONS:
Other: Pituitary function evaluation — Pituitary function evaluation performed at hospital discharge, 6 and 12 months
  * Thyroid-stimulating hormone, free T4 and T3
  * Follicle stimulating hormone, luteinizing hormone, estradiol, bioavailable testosterone
  * Adrenocorticotropic hormone stimulation test
  * Glucagon test (growth hormone deficit)
  Risk factors evaluation of pituitary dysfunction
  * Demographic data
  * Daily data (clinical exam, secondary brain injuries)
  * Hormone levels on day 1, 3 and 7
  * Biomarkers on day 1, 3 and 7
  * Brain CT-Scan on day 1
  * Pituitary MRI on day 7
  Outcome measures at 6 and 12 months
  * Neurological recovery (GOSe)
  * Independent functioning (FIM)
  * Quality of life (EQ-5D-5L)
  * Life satisfaction (LISAT-11)
  * Depression (PHQ-9)

SUMMARY:
Damage to the pituitary gland is a frequently overlooked but potentially important complication of traumatic brain injury (TBI). Disorders of the pituitary gland can cause dysfunction of the thyroid, adrenals, ovaries and testes. These disorders may occur immediately or several months after TBI, may delay recovery and may have a significant negative impact on quality of life. TBI is the leading cause of disability and major permanent functional impairment among adults under 45 years of age. Hormonal deficits may contribute to common symptoms experienced by TBI survivors such as fatigue, poor concentration, depression and low exercise capacity. However, the association between hormonal deficits and disability remains uncertain. The primary objective of this pilot study is to assess the feasibility of a larger study that will evaluate the impact of pituitary disorders on neurological disability and functional recovery. The results of this study will provide key findings in the impact of pituitary disorders following TBI, which is a mandatory step prior testing the effect of hormonal replacement therapy in this population in costly clinical trials. If no relationship between pituitary disorders and disability is observed, the investigators' findings will prevent unnecessary, time-consuming and costly hormonal screening and will discourage potentially harmful hormonal therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥ 18 years old)
* Severe or moderate blunt TBI admitted to the ICU with a Glasgow Coma Scale ≤ 12 following initial resuscitation

Exclusion Criteria:

* Previously diagnosed or suspected pituitary disorder or disease
* Pregnant or lactating woman
* Penetrating TBI
* Solid malignancy with life expectation <12 months
* Liver Cirrhosis Child C
* Chronic Heart Failure (New York Heart Association class IV)
* End-stage chronic respiratory disease (O2 dependent)
* End-stage renal disease (chronic dialysis or to be expected)
* Neurological conditions influencing functional status (e.g. spinal cord injury, neuromuscular disease, dementia, prior TBI or stroke)
* No fixed address
* Physician refusal
* Brain death
* Unable to return to the study center to attend the follow-up visits
* Admission to the Intensive Care Unit of the participating center > 24 hours after TBI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2015-03; Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Adherence to the Protocol | 12 months
  Percentage of participants who underwent pituitary function evaluation and outcome measures as detailed in the Assigned Interventions section
Enrollment Rate | 12 months
  Number of patients recruited per month per site

SECONDARY OUTCOMES:
Neurological Recovery | 12 months
  Glasgow Outcome Scale Extended (GOSe)
Quality of life | 12 months
  EuroQuol - EQ-5D-5L questionnaire
Independent functioning | 12 months
  Functional Independence Measure (FIM) questionnaire
Depression | 12 months
  Patient Health Questionnaire (PHQ-9)
Life satisfaction | 12 months
  Life Satisfaction Questionnaire (LISAT)
Secondary hypothyroidism | 12 months
Secondary hypogonadism | 12 months
Secondary adrenal insufficiency | 12 months
Growth hormone deficit | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: François Lauzier, MD MSc FRCPC, Principal Investigator — CHU de Quebec Research Center
Locations (5):
- Canada (5):
  - The Ottawa Hospital, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Hôpital du Sacré-Coeur de Montréal, Montreal, Quebec
  - CHU de Québec - Hôpital de l'Enfant-Jésus, Québec, Quebec
  - CHU de Sherbrooke - Hôpital Fleurimont, Sherbrooke, Quebec

REFERENCES:
- [Background] Lauzier F, Turgeon AF, Boutin A, Shemilt M, Cote I, Lachance O, Archambault PM, Lamontagne F, Moore L, Bernard F, Gagnon C, Cook D. Clinical outcomes, predictors, and prevalence of anterior pituitary disorders following traumatic brain injury: a systematic review. Crit Care Med. 2014 Mar;42(3):712-21. doi: 10.1097/CCM.0000000000000046. PMID 24247474
- See also: Related Info — http://www.ccctg.ca